CLINICAL TRIAL: NCT07194486
Title: Perceptions of Medical Students Toward Health Policy Education and Engagement in Policy Roles, Sudan 2025
Status: Completed | Type: Observational
Sponsor: Research and Publication office (Other)
Responsible Party: Sponsor
Other Study IDs: 24007
Record Dates: First submitted 2025-02-06; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-02

CONDITIONS: Perceptions of Health Policy Education; Engagement in Policy Roles
Keywords: Health Policy; Medical students; Awareness; Sudan

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study assesses medical students' perceptions of health policy education, their readiness for policy roles, and barriers to participation. Findings will highlight gaps and guide curriculum improvements in Sudan.

DETAILED DESCRIPTION:
This study aims to assess medical students' perceptions and knowledge regarding health policy education in undergraduate medical curricula. It seeks to evaluate their awareness and understanding of health policy concepts, assess the adequacy of health policy education, identify barriers to effective learning and participation, and explore students' interest and readiness to engage in policy-making. The findings will help identify gaps, strengths, and areas for improvement, offering valuable insights for curriculum development to enhance medical education outcomes in Sudan.

ELIGIBILITY:
Inclusion Criteria:

* All medical students enrolled in an accredited medical program at the time of the data collection.

Exclusion Criteria:

* Non medical students
* Postgraduates
* Student in foreign universities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All medical students in accredited medical universities.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Medical students perception of health policy education | Jan _ Mar 2025

SECONDARY OUTCOMES:
Exposure to formal education on health policy | Jan - Mar 2025
Confidence in applying policy concepts | Jan -Mar 2025
Satisfaction with current education | Jan - Mar 2025
Interest in engagement in policy roles | Jan - Mar 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Research and publication office, Khartoum, Omdurman, Sudan

IPD SHARING:
Plan to Share IPD: No